CLINICAL TRIAL: NCT00892476
Title: Prevention of Myopia of Prematurity by Calcium Supplementation in a Randomized Controlled Pilot Trial
Brief Title: Prevention of Myopia of Prematurity by Calcium Supplementation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F010613009
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2010-07

CONDITIONS: Myopia
Keywords: myopia; calcium supplementation; prematurity
MeSH Terms: conditions — Myopia; Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Infants receive supplemental calcium in their 24 cal/oz formula or fortified breast milk.
  Interventions: Dietary Supplement: Calcium Supplementation
- 2 (Active Comparator): Infants will receive fortified breast milk or 24 cal/oz formula
  Interventions: Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Calcium Supplementation — Ca-gluconate powder (molar weight 430.4 g) will be measured with household measuring spoons and added to the feeding mixtures as follows:
  Amount of feeding Actual Weight < 1000 g Actual Weight < 1000 g
  25 ml ¼ tsp 1/8 tsp
  50 ml ½ tsp ¼ tsp
  100 ml 1 tsp ½ tsp
  200 ml 2 tsp 1 tsp
  Other Names: USP grade Calcium gluconate powder from Sigma Chemical Company (Cat # C-8231, St. Louis, MO)
  Arms: 1
Other: Standard of Care — Infants are feed breast milk with fortifier or 24 cal/oz formula per standard of care
  Arms: 2

SUMMARY:
The purpose of this study is to determine if supplementation of calcium by the enteral route (gut feeding) to extremely low birth weight infants will lead to less myopia (nearsightedness) at 6-12 months postnatal age.

Secondly, the study will determine if calcium supplementation is well tolerated, if it reduces the molding of these premature infants' heads, and if it decreases myopia at the 18-22 month postnatal age visit.

DETAILED DESCRIPTION:
All infants admitted meeting the 401-1000gm birthweight and less than 14 day of age entry criteria will be screened for entry into the study. Infants may be excluded for the following: Major congenital malformations, including complex congenital heart disease (except open ductus arteriosus, atrial and ventricular septal defects), pulmonary malformations, bowel or anal stenosis or atresia, renal dysplasias, chromosomal anomalies, hydrops fetalis, bowel perforation or necrotizing enterocolitis stage 2A or greater before randomization.

Written informed consent of one parent or legal guardian must be obtained. The infants are randomized to receive unsupplemented feedings of breast milk or formula, or feedings supplemented with Ca-gluconate as outlined below.

Randomization will be stratified into the following groups: 401-750 g and 751-1000 g and performed according to a balanced block scheme with variable block size (2-6) using sealed opaque envelopes.

Total parenteral nutrition is given by nursery unit standards. Infant positioning is done by nursery unit standards.

Feeding mixtures:

Supplementation is started when enteral feeding amounts to 100 ml/kg. At that time, fortification is also introduced in infants receiving breast milk. Fortified human milk or 24 cal/oz formula, e.g. Similac Special Care 24 (SSC24), is used in all participating infants. Human milk is fortified with 1 pk Enfamil human milk fortifier per 25 ml (BMHMF).

Control group: Fortified human milk or 24 cal/oz formula. Supplemented group: Ca-gluconate powder (molar weight 430.4 g) will be measured with household measuring spoons (e.g. Rubbermaid (R)) and added to the feeding mixtures.

One eye exam will be performed at 6-12 months during routine follow-up visit. A second eye exam will be performed at 18-2 months during a follow-up visit which is part of the NICHD newborn follow-up clinic. Head measurements, specifically, front-to-back and side-to-side will be measured at randomization, 36 weeks postmenstrual age or discharge, whichever occurs first, and during the follow up visits. Urinalysis will be collected weekly.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a birthweight of 401 - 1000 g and postnatal age less than 14 days

Exclusion Criteria:

* Major congenital malformations including

  * complex congenital heart disease (except open ductus arteriosus, atrial and ventricular septal defects)
  * pulmonary malformations
  * bowel or anal stenosis or atresia
  * renal dysplasias
  * chromosomal anomalies
  * hydrops fetalis
  * bowel perforation or necrotizing enterocolitis stage 2A or greater before randomization.

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2002-02; Primary Completion 2004-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Supplementation of Ca by the enteral route to ELBW infants will lead to an increased cycloplegic refraction at 6-12 months postnatal age. | 6-12 months postnatal age

SECONDARY OUTCOMES:
Supplementation of Ca will lead to increased cycloplegic refraction at 18-22 months corrected age. | 18-22 months corrected age
Supplementation of Ca will lead to an increased cycloplegic refraction at 6-12 months postnatal age and at 18-22 months corrected age in infants who had no abdominal surgery or prolonged feeding intolerance | 6 months postnatal age to 18-22 months corrected age
Supplementation of Ca will reduce the dolichocephalic deformation of the infants' heads as measured by the FOD/BPD index. | 18-22 months corrected age
Supplementation of Ca will reduce the incidence of fractures. | birth to discharge
Supplementation of Ca will not increase the incidence of NEC stage 2A or greater. | birth to discharge
Supplementation of Ca will not increase the incidence of feeding intolerance. | birth to discharge
Supplementation of Ca is not associated with a change in the incidence of ROP. | birth to full vascularization of the retina
Supplementation of Ca will increase bone mineral density at 36 weeks postmenstrual age (only relevant if measurement is available). | 36 weeks postmenstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Carlo, MD, Principal Investigator — University of Alabama at Birmingham

REFERENCES:
- [Derived] Carroll WF, Fabres J, Nagy TR, Frazier M, Roane C, Pohlandt F, Carlo WA, Thome UH. Results of extremely-low-birth-weight infants randomized to receive extra enteral calcium supply. J Pediatr Gastroenterol Nutr. 2011 Sep;53(3):339-45. doi: 10.1097/MPG.0b013e3182187ecd. PMID 21865980